CLINICAL TRIAL: NCT05165186
Title: Care Planning for a Loved One With Dementia: Knowledge, Preparing for Decisions, and Emotions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Bradford Clark Dickerson, M.D., Director, Frontotemporal Disorders Unit and Laboratory of Neuroimaging, Massachusetts General Hospital, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2021P001869; 5R01AG061968-03 (NIH)
Record Dates: First submitted 2021-12-07; First posted 2021-12-21 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Dementia; Dementia Frontotemporal; Dementia Alzheimers; Dementia, Mild; Dementia Moderate; Dementia Severe; Caregiver Burnout; Caregiver Stress Syndrome
Keywords: Caregiving; Dementia; Frontotemporal Dementia (FTD); Caregiver Burden
MeSH Terms: conditions — Dementia; Pick Disease of the Brain; Alzheimer Disease; Lymphoma, Follicular; Caregiver Burden; Frontotemporal Dementia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video Intervention Arm (Experimental): For participants randomized to the video intervention arm, participants will be shown two videos about Advanced Care Planning, and then they will be asked questions regarding the usefulness of the video and their comfort with the video
  Interventions: Other: Video Intervention Arm
- Control Arm (No Intervention): For participants randomized to the control group arm, participants will review an informational sheet, which covers the same information as the videos shown to the intervention arm.

INTERVENTIONS:
Other: Video Intervention Arm — For participants randomized to the video intervention arm, participants will be shown two videos about Advanced Care Planning, and then they will be asked questions regarding the usefulness of the video and their comfort with the video.
  Arms: Video Intervention Arm

SUMMARY:
The overall objective of this study is to compare knowledge, decisional conflict, preferences, and caregiver burden over time caregivers of Alzheimer's Disease and Related Dementias (ADRD) patients by comparing the effectiveness of a video decision aid intervention and enhanced usual care.

DETAILED DESCRIPTION:
The investigators will conduct a randomized controlled trial in 150 caregivers of patients with ADRD, who will be randomized to either the video (intervention) or enhanced usual care (informational sheet, control). The intervention group will use the suite of video decision aids. Caregivers in the control group will review the informational sheet, which covers the same information.

Data collection is estimated to take no longer than an hour and will be conducted after the scheduled visit at the Massachusetts General Hospital Memory Disorders Unit (MGH MDU) clinic. The relatively brief interviewing time (30 minutes) in which the survey is conducted should assure completion of the interview without burdening participants. The investigators do not foresee the additional time to complete the survey to be a barrier to successful recruitment and completion of the protocol. Participants will be provided written copies of the questions in order to follow along during the face-to-face interviews.

The research assistant (RA) will collect baseline data, randomize caregivers to either the video or control arm via concealed envelopes, and administer the intervention. After this baseline interview and randomization, the RA will collect the remaining outcomes data regarding knowledge, preferences, decisional uncertainty, and caregiver burden from the caregiver. For those participants randomized to the video intervention, they will also be asked questions regarding the usefulness of the video and their comfort with the video. All caregivers will be given a website link to access the videos shown from their home. As the investigators have done in prior studies, the investigators will contact by telephone caregivers at 3 and 6 months to assess their caregiver burden at that time. Fidelity of the video intervention during the in-person survey and remotely at home will be tracked via a video website link that documents show-rates (date and time video accessed) as well as play-through rates (was the video watched to completion).

ELIGIBILITY:
Inclusion Criteria:

* All participants must be age 18 or older.
* Participants must be able to speak and understand English.
* Participants must be a caregiver of someone with Alzheimer's Disease, frontotemporal dementia, or a related dementia
* Participants should be able to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information (PHI) in accordance with national and local participant privacy regulations.

Exclusion Criteria:

* Participants who are not able to tolerate or perform the procedures or assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-04-13 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in percent correct and in response confidence on Knowledge of Advanced Dementia Questionnaire. | Baseline and immediately post-intervention
  The Knowledge of Advanced Dementia Questionnaire is a verbally administered self-reported instrument assessing knowledge with six true/false questions with a total possible score of 6 (1 point for each correct T/F), with high scores indicating better knowledge. A confidence rating scale with possible scores from 1 (not at all confident) to 5 (extremely confident).
  Change = (post Knowledge score - pre Knowledge score) Change = (post Confidence score - pre Confidence score)
Change from Baseline in percent correct and in response confidence on Knowledge of Goals of Care Questionnaire. | Baseline and immediately post-intervention
  The Knowledge of Goals of Care is a verbally administered self-reported instrument assessing knowledge with six true/false questions with a total possible score of 6 (1 point for each correct T/F), with high scores indicating better knowledge. A confidence rating scale with possible scores from 1 (not at all confident) to 5 (extremely confident).
  Change = (post Knowledge score - pre Knowledge score) Change = (post Confidence score - pre Confidence score)
Change and Retention of Change in Advanced Care Planning (ACP) Engagement Survey | Baseline and immediately post-intervention Post-intervention and 3 Month Follow Up Post Intervention and 6 Month Follow Up
  The ACP Engagement Survey is a self-reported instrument assessing confidence and readiness for ACP activities. Possible scores range from 1 (Not at all) to 5 (Extremely).
  Change = (Post intervention score - baseline score) Retention = (3 Month Follow Up - Post Intervention) Retention = (6 Month Follow Up - Post Intervention)

SECONDARY OUTCOMES:
Change and Retention of Change in Decisional Conflict Scale | Baseline and immediately post-intervention Post-intervention and 3 Month Follow Up Post Intervention and 6 Month Follow Up
  The Decisional Conflict Scale is a validated, self-reported instrument assessing 5 dimensions of decision-making feelings (uncertain, uninformed, unclear about values, unsupported; ineffective decision making). Possible scores range from 1 (strongly disagree) to 5 (strongly agree).
  Change = (Post intervention score - baseline score) Retention = (3 Month Follow Up - Post Intervention) Retention = (6 Month Follow Up - Post Intervention)
Response Rate and Retention of Response Rate for Limited Medical Care and Comfort Care | Baseline and immediately post-intervention Post-intervention and 3 Month Follow Up Post Intervention and 6 Month Follow Up
  The ACP Preferences Survey is a self-reported instrument asking a one multiple choice question with 3 options; Life Prolonging Care, Limited Medical Care and Comfort Care.
  Change = (Post intervention response rate - baseline response rate) Retention = (3 Month Follow Up response rate - Post Intervention response rate) Retention = (6 Month Follow Up response rate - Post Intervention response rate)
Response Rate for Advanced Care Planning (ACP) Documents Survey | Baseline and Month 3 Follow Up Baseline and Month 6 Follow Up
  The ACP Documents Survey is a self-reported instrument asking 3 yes/no/unsure questions assessing the completion of ACP documents with a total possible score of 3 (1 point for each yes answer). A higher score indicates a higher amount of documents completed.
  Change = (3 month follow up score - baseline score) Change = (6 month follow up score - baseline score)
Response Rate of Satisfaction Survey on Video Rating Survey post-intervention | Immediately post-intervention
  Responses from the Video Rating Survey, a self-reported instrument asking 5 questions assessing perception of ACP Video: Goals of Care: Advanced Dementia. Possible scores range from 1 (strongly disagree) to 5 (strongly agree) for knowledge, comfort, desire to learn more and recommend to others with a higher summary score indicating a positive response except for comfort, where a higher response indicating more discomfort. Importance to learn about this topic was measured on a 5-point scale; 1 (Not at all important) to 5 (Very Important) with a higher summary score indicating higher importance.

OTHER OUTCOMES:
Change from Baseline self-report measure of affect to post intervention self-report measure of affect | Baseline and immediately post-intervention
  The PANAS is a validated self-report instrument assessing affect. Possible answers range from 1 (Very slightly or not at all) to 5 (Extremely) The total score is calculated by finding the sum of the 10 positive items and then the 10 negative items. Scores range from 10 - 50 for both sets of items. For the total positive score, a higher score indicates more of a positive affect. For the total negative score, a lower score indicates less of a negative affect.
  Change = (Post-intervention - Baseline)

CONTACTS AND LOCATIONS:
Overall Officials: Brad C Dickerson, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share individual participant data that underlie the results reported in each published article, after deidentification
Supporting Information: Study Protocol
Time Frame: After publication of article
Access Criteria: Researchers who provide a methodologically sound proposal